CLINICAL TRIAL: NCT06332391
Title: A New Pacing Approach for Cardiac Conditioning and Enhanced Cardioprotection
Brief Title: Paced Heart Rate Acceleration for Cardiac Conditioning
Acronym: HeartExcel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Denice Hodgson-Zingman, MD (Other)
Collaborators: The Cleveland Clinic (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Denice Hodgson-Zingman, MD, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202308349; R01HL168752 (NIH)
Record Dates: First submitted 2023-11-27; First posted 2024-03-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure, Systolic
Keywords: heart failure; exercise; heart rate; implantable defibrillator; cardiac conditioning; exercise tolerance; pacing; cardiac output; quality of life; walking distance
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective, single blinded, randomized, controlled trial. Randomization to intervention versus sham groups in a 1:1 ratio.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Subjects and outcomes assessors are blinded to study group (intervention vs. sham) but investigator is not. During intervention vs. sham, subjects do not have access to vital sign data and sham procedures follow intervention procedures exactly with the exception that no change in pacing rate is delivered. A blinding questionnaire is given to subjects to assess adequacy of blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise-similar cardiac pacing (Experimental): Atrial pacing to replicate exercise heart rate envelope once daily, 3 days per week, over 6 weeks while symptoms and vital signs are monitored and outcome measures assessed.
  Interventions: Device: Exercise-similar cardiac pacing
- Sham cardiac pacing (Sham Comparator): Sham pacing to replicate exercise heart rate envelope once daily, 3 days per week, over 6 weeks while symptoms and vital signs are monitored and outcome measures assessed.
  Interventions: Device: Sham cardiac pacing

INTERVENTIONS:
Device: Exercise-similar cardiac pacing — Cardiac pacing using subjects already-implanted cardioverter defibrillator to reproduced exercise heart rate envelope.
  Arms: Exercise-similar cardiac pacing
Device: Sham cardiac pacing — Simulated (rates selected using programmer but not initiated) cardiac pacing using subjects already-implanted cardioverter defibrillator to reproduced exercise heart rate envelope.
  Arms: Sham cardiac pacing

SUMMARY:
A clinical trial of exercise-similar heart rate acceleration delivered via cardiac pacing vs. sham intervention in subjects at rest will be performed. The study population comprises subjects with guideline-directed medically managed left ventricular dysfunction due to ischemic or non-ischemic cardiomyopathy and an existing implantable cardioverter defibrillator or biventricular implantable cardioverter defibrillator. The purpose of the study is to understand how the heart rate pattern of exercise contributes to the considerable cardiac conditioning effects of exercise and estimate whether the pacing approach may have translational clinical applicability. Fifty-two subjects will be randomized, single-blinded, to either the pacing intervention or a sham intervention which they will receive once daily, 3 days/week for 6 weeks. Baseline symptoms and clinical test results will be compared to the same measures at 2 weeks, 4 weeks and 6 weeks of intervention/sham and at 3 months and one-year post-intervention. The primary endpoint will be the change in left ventricular ejection fraction from baseline in intervention vs. sham groups (mixed effects linear regression with time and treatment arm as fixed effects and pre-specified covariates of sex and cardiomyopathy type as random effects). Secondary endpoints will include changes in quality of life, 6-minute walk distance, cardiopulmonary exercise test (CPET) measures, daily activity and major adverse cardiac events (MACE) at 3 and 12 months between pacing and sham groups. A "dose-response" analysis of outcomes at 2, 4, and 6 weeks of the intervention vs. sham compared with baseline will be performed.

DETAILED DESCRIPTION:
Subjects and protocol: This is a phase II randomized, controlled, prospective clinical trial in subjects with systolic heart failure. It is designed to assess the effect on symptoms, functional, structural, and medical outcomes in response to an atrial paced reproduction of the heart rate exercise pattern delivered regularly over a 6-week period. A single center (University of Iowa) will execute the intervention/sham and subject testing. A separate center (Cleveland Clinic) will perform statistical analysis of deidentified data. Fifty-two subjects will be randomized 1:1 by computer generated code to either the intervention (pacing) arm or the sham arm. The subject, but not researcher, will be blinded to randomization status (single-blind). Analysis of data will be performed in a blinded fashion. Within 2 weeks prior to initiation of pacing vs. sham interventions, baseline testing will be performed including collection and storage of plasma, testing for blood urea nitrogen (BUN), creatinine, N-terminal pro-b-type natriuretic peptide (NT-proBNP), echocardiographic left ventricular (LV) dimensions, left ventricular ejection fraction (LVEF), and quality of life/symptoms by both the Minnesota Living with Heart Failure (MLHF) and the Kansas City Cardiomyopathy Questionnaire (KCCQ), designed for assessment of symptoms over 1 month and 2 week windows, respectively, distance on 6-minute walk, 1 week of pacing device accelerometer-derived activity measures, wearable activity monitor measures, and cardiopulmonary exercise test (CPET) for determination of metabolic equivalents (METs), maximum oxygen consumption (VO2max) and anaerobic threshold (AT) estimated noninvasively, using the rapid incremental exercise test. In addition, starting 1 week prior and continuing through 1 month after the pacing vs. sham intervention, each subject will be provided a wearable activity monitor and their daily activity analyzed as a cofactor. At the end of 2, 4 and 6 weeks of pacing/sham, as well as 3 and 12 months after the intervention, the same outcome measures as at baseline will be collected as well as major adverse cardiovascular events (MACE), weight, medications, and arrhythmias recorded on the subject's implantable cardioverter defibrillator (ICD) or biventricular ICD (BiV/ICD). At the end of the pace/sham period, subject blinding will be assessed by asking subjects if they believe they were in pace or sham group. Collected plasma will be saved for metabolomic testing in year 5 to correlate with findings in mouse models. Outcomes: All tests result analyses will be done by 2 independent clinicians, qualified in specific areas, blinded to the randomization. A reviewer who analyzes a testing parameter will analyze the same parameter for all subjects. Variability between reviewers will be analyzed. The primary endpoint will be change in left ventricular ejection fraction (LVEF) from baseline. Secondary endpoints will include quality of life (QOL) by MLHF score, 6-min walk distance, CPET (including VO2max, metabolic equivalents (METs) achieved, peak power output, total exercise time), daily activity change from baseline and MACE at 3 and 12 months between pacing and sham groups. A "dose-response" analysis of outcomes at 2, 4, and 6 weeks of the intervention vs. sham compared with baseline will be performed. Durability analysis of response at 3 and 12 months will be performed.

The data from all subjects completing at least one pacing vs. sham session will undergo analysis for measures of tolerability (symptoms, maximum achieved pacing rate, appearance of arrhythmias, changes in vital signs and bioimpedance cardiac output) with respect to age, sex, degree, type of cardiomyopathy (ischemic vs. non-ischemic), left ventricular function, NT-proBNP, NHYA class, baseline oxygen consumption (VO2), baseline exertional tolerance, baseline physical activity level as assessed by the ICD of BiV/ICD accelerometer and wearable activity watch, autonomic function as defined by heart rate variability derived from electrocardiogram (ECG) and stored ICD or BiV/ICD data. Hospitalizations, deaths, or other adverse outcomes will similarly be analyzed with respect to baseline data and procedural data such as maximum achieved pacing rate.

For those subjects completing the intervention/sham and follow up visits, the primary endpoint of change in left ventricular ejection fraction will be analyzed. Secondary endpoints will include changes in functional capacity, particularly 6-minute walk, and quality of life indicators as well as MACE with respect to the above study variables.

Descriptive statistics will be used to summarize participant demographic and clinical characteristics at baseline. Categorical variables will be compared using Chi squared tests. For continuous variables, to relax the strict requirement of normality, non-parametric methods for unadjusted comparison will be used (Wilcoxon rank-sum test, also known as the Mann-Whitney two-sample statistic, for comparison of two independent samples. Wilcoxon matched pairs signed-rank test will be used for paired comparisons). For the primary endpoint analysis, a mixed-effects linear regression model will be used to compare the two study arms on the primary outcome of LVEF, with time (2, 4, and 6 wks) and treatment arm (intervention vs. sham) included as fixed effects, and pre-specified covariates of sex (binary male/female) and cardiomyopathy type (binary ischemic/non-ischemic) as random effects. Both stratified randomization by sex and cardiomyopathy type, as well as adjustment for these covariates in the analysis, will be performed. Although often only one or the other technique is sufficient, both are performed here given the well-known confounding effects of sex and cardiomyopathy types in heart failure trials and a desire to be highly rigorous in this regard. An intercept for time of treatment or sham (2, 4, 6 wks) will be included. The significance criteria for the model coefficient corresponding to treatment will be .025 with a one-sided 97.5% confidence interval. Analyses will be conducted on an "intention-to-treat" basis. Estimates and confidence intervals of effect sizes and standard deviation of outcome measures will be presented. Pre-specified subgroup analyses will probe for treatment effect heterogeneity in outcomes based on sex and ischemic cardiomyopathy vs. nonischemic cardiomyopathy. Secondary endpoints will be analyzed in a fashion similar to the primary endpoint analysis. Due to the controlled environment, missing data are expected to be very rare. If such exists, patterns will be evaluated, and multiple imputation performed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female sex
* Age 18 years or greater
* Available transportation for study visits
* Left ventricular ejection fraction < or = 40% despite at least 3 months guideline-directed medial therapy
* NYHA class II-III heart failure symptoms
* Atrial-lead inclusive implantable cardioverter defibrillator or biventricular defibrillator in place > 3 months
* Intrinsic or biventricular paced QRS duration of <= 120 milliseconds

Exclusion Criteria:

* Age < 18 years
* Inability to ambulate safely
* Congenital or primary valve disease
* Ongoing (not suppressed) atrial arrhythmias
* Left ventricular thrombus
* Severe peripheral arterial disease that limits mobility
* Hospital admission for life-threatening condition (e.g. heart failure, stroke) in the past 3 months
* Major surgery in the past 3 months or anticipated during the period of study
* Ventricular pacing indication in the absence of biventricular pacing
* Life expectancy < 1 year
* Hemodialysis
* Hematocrit < 30%
* Severe chronic lung disease that limits activity or requires oxygen
* Pregnancy
* Implantable cardioverter defibrillator battery longevity < 1 year
* Vulnerable populations such as prisoners and institutionalized individuals

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction by echocardiogram | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  The change in left ventricular ejection fraction from baseline as determined by echocardiography

SECONDARY OUTCOMES:
Quality of Life score on the Minnesota Living with Heart Failure questionnaire | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  Numerical score based on a subject's subjective symptoms and functional status
Quality of Life score on the Kansas City Cardiomyopathy Questionnaire | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  Numerical score based on a subject's subjective symptoms and functional status
6-minute walk distance | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  Distance on a standard 6-minute walk measured in meters
Cardiopulmonary exercise test maximum oxygen consumption | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  V02max (maximum milliliters of oxygen consumed per kilogram of body weight per minute)
Cardiopulmonary exercise test metabolic equivalents achieved | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  metabolic equivalents (METs)
Cardiopulmonary exercise test peak power output achieved | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  peak power output (watts/kilogram)
Cardiopulmonary exercise test total exercise time | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  total exercise time (minutes)
daily minutes of sedentary activity | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  CamNtech motion watch 8 average daily minutes of activity in the sedentary range
daily minutes of low activity | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  CamNtech motion watch 8 average daily minutes of activity in the low range
daily minutes of moderate activity | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  CamNtech motion watch 8 average daily minutes of activity in the moderate range
daily minutes of vigorous activity | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  CamNtech motion watch 8 average daily minutes of activity in the vigours range
major adverse cardiac events | at baseline versus 2 weeks, 4 weeks, 6 weeks from start of intervention/sham and at 3 months and 12 months after completion of intervention vs. sham.
  MACE
symptom score during the intervention/sham procedure | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  An aggregate score of a subject's subjective report of shortness of breath, chest pain, palpitations, lightheadedness, each on a scale of 0-10. Minimum score 0, maximum score 40.
maximum achieved pacing rate during the intervention/sham procedure | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  measured in beats/minute
presence of significant arrhythmia during the intervention/sham procedure | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  binary outcome of 0 (no such arrhythmia) versus 1 (presence of a significant arrhythmia) during each episode of pacing. A significant arrhythmia refers to either subject-reported symptoms during the arrhythmia, or a change in systolic blood pressure of 20 mmHg from that immediately before the onset of the arrhythmia, or an arrhythmia requiring intervention to terminate.
vital signs - systolic blood pressure during the intervention/sham procedure | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  maximum change in systolic blood pressure (millimeters of mercury) during the intervention/sham period versus the baseline blood pressure immediately before initiation of intervention/sham procedure as measured by plethysmography (standard inflatable blood pressure cuff).
vital signs - oxygen saturation in the blood during the intervention/sham procedure | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  maximum change in blood oxygen saturation (measured as % saturation) during the intervention/sham period versus the baseline immediately before initiation of intervention/sham procedure as measured by pulse oximeter.
tolerability - vital signs - cardiac output | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  maximum change in cardiac output during the intervention/sham period versus the baseline immediately before initiation of intervention/sham procedure as measured by NICaS bioimpedance device.
vital signs - cardiac output during the intervention/sham procedure | at each intervention/sham procedure - these occur 3 days per week for 6 weeks at the beginning of the study
  maximum change in cardiac output (liters/minute) during the intervention/sham period versus the baseline immediately before initiation of intervention/sham procedure as measured by NICaS bioimpedance device.

CONTACTS AND LOCATIONS:
Overall Officials: Denice Hodgson-Zingman, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States